CLINICAL TRIAL: NCT05713825
Title: Multidimensional Evaluation of Patients With Ruptured or Unruptured Cerebral Aneurysm Undergoing Endovascular or Surgical Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Alexandre Andrea, MD MSc, Principal Investigator, Neuroradiologist, MD MSc, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 3583
Record Dates: First submitted 2023-01-26; First posted 2023-02-06 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Cerebral Aneurysm
MeSH Terms: conditions — Intracranial Aneurysm | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Endovascular embolization or surgery — * Endovascular embolization may be done with coils, remodeling technique (coils and balloon), stent and coils, flow-diverter, endosaccular devices. The access is through the femoral or radial artery.
  * Surgery is considered the standard neurosurgical procedure of aneurysm clipping.

SUMMARY:
Cerebral aneurysms are common changes in intracranial angioarchitecture. Unruptured aneurysms are increasingly identified thanks to the imaging techniques used in daily clinical practice. Since bleeding remains a highly dramatic event burdened by significant morbidity-mortality (about 50%), endovascular therapy, in combination with classic surgical therapy, is an essential element in contemporary medicine.

Endovascular and surgical treatment represent the standard of care. The rationale of this study is to identify clinical and radiological characteristics, mainly neuro-radiological ones, not fully explored in previous studies, which can help predict the outcome of patients affected by cerebral aneurysm.

The study will have the characteristics of a retrospective study on patients with cerebral aneurysm treated at our center from 1 January 2015 to 31 December 2023.

Objective of the study is the multidimensional evaluation in patients with cerebral aneurysms, ruptured and unruptured, undergoing an endovascular embolization procedure or surgical treatment.

DETAILED DESCRIPTION:
Cerebral aneurysmal disease affects 2-5% of the world population, with 0.7-1.9% of cases of rupture resulting in subarachnoid hemorrhage (SAH). The most affected age group is wide - from 30 to 60 years - with a ratio between male and female gender equal to 1.6.

SAH accounts for approximately 5% of strokes and is burdened by high mortality and disability rates; in this particular situation, the patient is subjected in the shortest time possible to a clinical-anamnestic framework, to evaluate the severity of the clinical picture and quantify it through the use of the Hunt & Hess scale, which is followed by the direct tomographic examination, to evaluate the extent of the lesions.

Recently, numerous developments have been observed in the treatment, elective or acute, of cerebral aneurysm, such as the introduction of new therapeutic devices, such as the flow diversion stent or "flow diverter".

The primary objective of the treatment of a cerebral aneurysm must be different on the basis of the type of lesion and the patient's clinical conditions: while, in fact, the treatment of a ruptured aneurysm has the primary aim of avoiding immediate rebleeding and facilitating treatment intensive, the goal of treatment of an unruptured aneurysm must be the achievement of a stable result, up to and including exclusion from the circulation.

Endovascular therapy has reached such prominence that, in most teams, the right of first refusal in the treatment of aneurysmal subarachnoid hemorrhage rests with the interventional neuroradiologist and no longer with the neurosurgeon.

The scientific literature is now rich in this regard, and in particular the two ISUIA (International Study of Unruptured Intracranial) trials and the ISAT (International Subarachnoid Aneurysm Trial ) are two points of reference in the management of intracranial aneurysms nowadays, focusing on endovascular treatment, especially in suitable anatomical conditions.

Although clinical trials and meta-analyses have dispelled any doubts about the validity/necessity of the therapies, the authors are convinced that there may be clinical and radiological characteristics, not fully explored in the aforementioned studies, which can help predict the outcome of these patients. The finding of these variables, if confirmed by subsequent trials aimed at the purpose, could in the future guide the selection of patients to undergo treatment as well as guide the choice of the best technique, endovascular or surgical in primis, to be applied according to the characteristics of each patient .

Therefore, it is the authors' intention to conduct a retrospective observational study with the aim of exploring the possible implication of new variables that can predict with sufficient accuracy the outcome of patients with ruptured and unruptured cerebral aneurysms; a possible positive response could be followed by a more structured clinical trial with which to derive the appropriate conclusions with greater methodological soundness.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* ruptured or unruptured cerebral aneurysm with consistent neurologic and radiologic evidence.
* CT without contrast medium and CT angiography, demonstrating the SAH and the aneurysm.
* Execution of an endovascular embolization procedure (which is indicated by a neurosurgeon and interventional neuroradiologist) or surgical treatment.

Exclusion Criteria:

* non-aneurysmal causes of SAH (example: AVMs, AVDs and trauma).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Given the purely descriptive nature of the primary objective, we do not proceed with the formal calculation of the sample size but a sample of N=500 patients is proposed.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-31 (Estimated); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Functional independence at 90 days assessed by Rankin scale (mRS). | 90 days
  A good clinical outcome will be defined as an modified Rankin Scale (mRS) score between 0 and 2 (mRS 0 identifies a patients with no symptoms, 6 identifies a dead patient).

SECONDARY OUTCOMES:
efficacy of endovascular treatment using the Raymond-Roy scale | at the end of the endovascular procedure
  Raymond-Roy scale:
  class I: complete obliteration class II: residual neck class III: residual aneurysm
90-day in-hospital mortality. | 90 days
  Any cause of death in patients treated for a cerebral aneurysm (considering endovascular or surgical procedures)
post-procedural symptomatic stroke/haemorrhage. | 48 hours after the procedure
  Any type of symptomatic ischemic or hemorrhagic event following endovascular or surgical procedures

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A.Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No